CLINICAL TRIAL: NCT04490031
Title: Randomized Control Study Evaluating Ketamine as Sedative Agent in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Evaluation of Ketamine as Sedative Agent in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: Hukm
Record Dates: First submitted 2020-03-24; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-03

CONDITIONS: Ketamine Adverse Reaction
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both the patients and surgeon will be blinded from knowing the sedative agent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Midazolam group (No Intervention): Standard sedation for ERCP in UKMMC
- Ketamine group (Experimental)
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — patient in Ketamine group will be given Ketamine as sedative agent
  Arms: Ketamine group

SUMMARY:
This is a study evaluating the usage of Ketamine as sedative agent in ERCP. The usage of Ketamine will be compared to the standard sedation in our center, which is Midazolam in combination with Pethidine as analgesia.

DETAILED DESCRIPTION:
This is a double blinded study whereby both the surgeons and patients are blinded from the sedative agent used. Patients admitted to UKMMC requiring ERCP will randomized into 2 groups after evaluating the inclusion and exclusion criteria. Patients will be divided into two arms, Midazolam and Ketamine group respectively. Before the initiation of the the scope, patient would be given specified dose of sedation accordingly. All the parameters and outcome would be measured during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizens of who is able to give valid consent
* Patient planned for ERCP (either emergency or elective)

Exclusion Criteria:

* Known hypersensitivity towards Ketamine or Midazolam
* Patient refusal to participate or unable to give consent
* Increased intracranial pressure, acute stroke (<3 months), intracranial haemorrhage (<3 months)
* Uncontrolled hypertension (BP>160/100) and tachycardia (Heart rate >120)
* Acute myocardial infarction, acute coronary syndrome (<3 months)
* Tachyarrythmia
* Pregnancy
* IVDU or substance abuse patient
* Patient with history of hallucination
* Child's Pugh Class C

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
depth of sedation | 1 hour
  based on Ramsay Sedation Scale, from a scale of 1-6.
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response The aim of sedation is a score of 3-4
completion rate | 1 hour
  to evaluate completion rate between Ketamine and Midazolam group

SECONDARY OUTCOMES:
Surgeon satisfaction score | within 4 hours after completion of ERCP
  subjective scoring of surgeon regarding overall experience of the ERCP from a score of 0-10.
  0- poor, 5- moderate, 10- excellent
Patient satisfaction score | within 4 hours after completion of ERCP
  subjective scoring of patients regarding overall experience of the ERCP from a score of 0-10.
  0- poor, 5- moderate, 10- excellent
evaluate the occurrence of hypertension, hypotension, bradycardia, tachycardia, hypoxia, respiratory rate abnormality, nausea, vomiting and emergence symptoms | 24 hours
  recording the adverse events of each sedation.
  1. Hypotension: defined as a systolic blood pressure drop greater than 20mmHg to a value less than 90mmHg
  2. Hypertension: defined as a systolic blood pressure increase greater than 20mmHg or to a value more than 140mmHg
  3. Bradycardia: defined as heart rate less than 50 after the initiation of sedation or decrease in heart rate more than 20 beats per minute
  4. Tachycardia: defined as heart rate more than 100 after the initiation of sedation or increase in heart rate more than 20 beats per minute
  5. Hypoxia: defined by oxygen saturation less than 95%
  6. Respiratory rate abnormality
  7. Nausea, vomiting, emergence symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chik, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre; Norma mohamad, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre; Zamri Zuhdi, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre; Azlanudin Azman, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre; Muhammad Hafiz Ismail, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- University Kebangsaan Malaysia Medical center, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No